CLINICAL TRIAL: NCT01034436
Title: Fatty Acid Quality and Overweight
Brief Title: Fatty Acid Quality and Overweight (FO-study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Stine Marie Ulven, Associate professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 6.2008.1368
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Weight Reduction and Insulin Sensitivity
MeSH Terms: conditions — Weight Loss; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low intake of ALA and triacylglycerols (Placebo Comparator): Sunflower oil
  Interventions: Dietary Supplement: fatty acid quality and overweight
- high intake of ALA and triacylglyceroles (Experimental): Canola and linseed oils
  Interventions: Dietary Supplement: fatty acid quality and overweight
- high intake of ALA and diacylglycerols (Experimental): Canola and linseed oils
  Interventions: Dietary Supplement: fatty acid quality and overweight

INTERVENTIONS:
Dietary Supplement: fatty acid quality and overweight — Duration 12 weeks

SUMMARY:
The purpose of this study is to study the health effects of fatty acid quality in healthy, overweight individuals.

ELIGIBILITY:
Inclusion Criteria:

* no use of medication, healthy, 27<BMI<40

Exclusion Criteria:

* pregnant and lactating women, chronic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Will intake of fat as diacylglycerols give weight reduction in overweight individuals? | baseline (0 weeks), 12 weeks

SECONDARY OUTCOMES:
Will a high intake of ALA involve reduced levels of inflammatory markers? | baseline (0 weeks), 12 weeks
Will a high intake of ALA involve changes in insulin sensitivity? | baseline (0 weeks), 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stine Marie Ulven, PhD, Study Chair — Oslo and Akershus University College
Locations (1):
- Akershus University College, Oslo, Lillestrom, Norway

REFERENCES:
- [Derived] Telle-Hansen VH, Christensen JJ, Formo GA, Holven KB, Ulven SM. A comprehensive metabolic profiling of the metabolically healthy obesity phenotype. Lipids Health Dis. 2020 May 9;19(1):90. doi: 10.1186/s12944-020-01273-z. PMID 32386512